CLINICAL TRIAL: NCT00145951
Title: Randomized Trial of a Motivational Interview Versus Brief Advice in Primary Care to Engage Mid-Late Adolescents With a Web-based Depression Prevention Intervention
Brief Title: Reducing the Risk of Developing Major Depression in Adolescents/Young Adults With Minor Depression/Depression Symptoms
Status: Terminated | Type: Observational
Why Stopped: Lost funding
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13798A
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Motivational Interviewing; Crisis Intervention; Primary Health Care

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (3):
- 1
- 2
- 3
  Interventions: Behavioral: motivational interviewing, brief advice in primary care

INTERVENTIONS:
Behavioral: motivational interviewing, brief advice in primary care — motivational interviewing, brief advice in primary care
  Groups: 3

SUMMARY:
The purpose of this research study is to assess the feasibility of a combined primary care/web-based depression prevention intervention. Primary care physicians (PCP) currently lack an alternative behaviorally-based approach to antidepressant medications for individuals with depression symptoms or minor depression, but who have not yet developed Major Depression.

The objective of this study is to compare the feasibility and efficacy of motivational interviewing (MI) versus brief advice in primary care to engage adolescents with a web-based depression prevention intervention.

DETAILED DESCRIPTION:
There is no population-based approach to prevent the onset of major depression in adolescence. Adolescents with current sub-threshold depression symptoms (not meeting criteria for major depression, 5 < symptoms including depressed mood, irritability or loss of pleasure), a personal history of a depressive episode in the past or with a family history of depressive disorders are at increased risk. Because most adolescents have regular contact with primary care physicians, the primary care clinics could provide a setting to disseminate evidence-based preventive approaches. We have developed a combined primary care/Web-based preventive intervention to reduce the risk of developing depressive disorders in adolescents and young adults by adapting interventions of demonstrated benefit in study settings to a primary care/Web-based format in collaboration with leading investigators in the field. The goal of this research program is to evaluate the feasibility and possible efficacy of an alternative delivery mechanism for evidence-based behavioral approaches to depression treatment and prevention that have already demonstrated benefit with face-to-face delivery in study settings. Each component this intervention will need to be carefully evaluated for acceptability, safety, feasibility and efficacy. The focus of this study is the primary care component.

ELIGIBILITY:
Inclusion criteria include:

* (1) age 14-18 years and
* (2) one risk factor for developing depression in the next two years: sub-clinical depressed mood (not meeting criteria of major depression),
* a family history of depression in a parent or sibling, or past personal history of depression or personal perception of risk depression and desire to participate

Exclusion Criteria:

* criteria include meeting criteria or undergoing active treatment for major depression (5 or more symptoms nearly every day with functional impairment, minor depression),
* bipolar disorder,
* panic disorder,
* conduct disorder,
* substance abuse or having suicidal ideation.
* Active treatment for depression is defined as receiving anti-depressant medication or counseling within one year of remission of symptoms from the most recent episode.
* Those who meet DSM-IV criteria for minor depression (3-4 symptoms) or who report significant functional impairment (very difficult or above on the Prime MD functional impairment scale) will be notified and offered a referral for an evaluation by a mental health specialist (and will be strongly encouraged to attend).
* Those with 1-2 symptoms of depression will also be offered evaluation and treatment from a mental health specialist. In each case, the primary care physician will be notified and the parents (if under the age of 19).

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Subjects are between the ages of 14-18 years and
  * have one risk factor for developing depression in the next two years:
  * sub-clinical depressed mood (not meeting criteria of major depression),
  * a family history of depression in a parent or sibling, or
  * past personal history of depression or personal perception of risk depression and desire to participate
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Voorhees, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States